CLINICAL TRIAL: NCT02563821
Title: Programmed Intermittent Epidural Bolus Versus Continuous Epidural Infusion for Third Trimester Medical Termination of Pregnancy Analgesia : a Randomized Study.
Brief Title: Programmed Intermittent Epidural Bolus Versus Continuous Epidural Infusion for Third Trimester Medical Termination of Pregnancy Analgesia : a Randomized Study. (PCEA-IMG)
Acronym: PCEA-IMG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: I14032 (PCEA-IMG)
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Anesthesia, Epidural
Keywords: Termination of pregancy; Third trimester; Programmed intermittent epidural bolus; Continuous epidural infusion; Epidural analgesia; Legally induced abortion
MeSH Terms: interventions — Levobupivacaine; Sufentanil; Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PCEA-DC (Active Comparator): Injection of a 2 mL initial epidural loading dose consisting of a blend (10 mL) of levobupivacaine 20 mg, sufentanil 10 µg to assure the absence of motor block and so exclude intrathecal placement of the epidural catheter.
  * Injection of the rest of the loading dose (8mL).
  * In this group the pump is programmed to deliver a continuous infusion at 10 mL /h consisting of levobupivacaine 0,573 mg/mL, sufentanil 0,37 µg/mL, clonidine 1,38 µg/ mL. Additional 5 mL patient-activated boluses will be allowed with a lockout interval of 10 minutes.
  * If the parturient feels she has inadequate analgesia after having activated the PCEA bolus twice in a thirty minutes period, an additional manual bolus of 6 mL of levobupivacaine 2,5 mg/mL will be administered until the Pain Visual Analog Scale (PVAS) is < 3/10.
  Interventions: Procedure: Patient Controlled Epidural Analgesia for third trimester termination of preganancy analgesia; Drug: Levobupivacaine; Drug: sufentanil; Drug: clonidine; Device: epidural catheter
- PCEA-BIP (Active Comparator): Injection of a 2 mL initial epidural loading dose consisting of a blend (10 mL) of levobupivacaine 20 mg, sufentanil 10 µg to assure the absence of motor block and so exclude intrathecal placement of the epidural catheter.
  * Injection of the rest of the loadind dose (8 mL)
  * In this group the pump is programmed to deliver automated mandatory boluses of 5 mL consisting of levobupivacaine 0,573 mg/mL, sufentanil 0,37 µg/mL, clonidine 1,38 µg/mL every 30 minutes. Additional 5 mL patient-activated boluses will be allowed with a lockout interval of 10 minutes.
  * If the parturient feels she has inadequate analgesia after having activated the PCEA bolus twice in a thirty minutes period, an additional manual bolus of 6 mL of levobupivacaine 2,5 mg/mL will be administered until the Pain Visual Analog Scale (PVAS) is < 3/10 (0 = no pain and 10 = insufferable pain).
  Interventions: Procedure: Patient Controlled Epidural Analgesia for third trimester termination of preganancy analgesia; Drug: Levobupivacaine; Drug: sufentanil; Drug: clonidine; Device: epidural catheter

INTERVENTIONS:
Procedure: Patient Controlled Epidural Analgesia for third trimester termination of preganancy analgesia
Drug: Levobupivacaine
Drug: sufentanil
Drug: clonidine
Device: epidural catheter

SUMMARY:
Background : Recently, delivery of local anaesthetics via Programmed Intermittent Epidural Bolus (PIEB) has been shown to improve labour epidural analgesia compared to delivery via Continuous Epidural Infusion (CEI).

Purpose : However, the superiority of PIEB compared to CEI has not been investigated for third trimester voluntary termination of pregnancy.

We hypothesized that PIEB administration would result in a better degree of satisfaction of the patients compared with CEI for third trimester legally induced abortion analgesia.

DETAILED DESCRIPTION:
Abstract : The recent technical advances in antenatal diagnosis have led to an increase number of legally induced abortion at the third trimester of pregnancy. Psychological pain is frequently associated to physical pain in these kinds of interventions. So anaesthetists are more and more involved in voluntary termination of pregnancy analgesia.

In France, Patient Controlled Epidural Analgesia (PCEA) with CEI mode is usually used for voluntary termination of pregnancy analgesia. But recent studies have shown that PIEB mode as compared to CEI mode increases maternal satisfaction during labour. This may be attributed to a more extensive spread of epidural solution when delivered as a bolus rather than continuous infusion.

Few trials have been interested in investigating the best mode of PCEA for legally induced abortion analgesia.

This study includes women who undergo voluntary third semester termination of pregnancy. Patients are randomized to PIEB or CEI for pain analgesia. In this randomized, double-blind study, the investigators assess the degree of satisfaction of the patients (primary outcome), the incidence of motor block, total drug consumption and adverse events (secondary outcomes) between the two study groups.

The different values are collected during the intervention on a specific paper for each patient and the degree of satisfaction is reported on this paper just before the patient leaves the birth room (approximatively 2 hours after the expulsion).

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* ASA 1 or 2 (healthy women)
* pregnancy at third trimester
* willingness of voluntary interrupt the pregnancy
* women affiliated to french health social system
* written informed consent from every patient

Exclusion Criteria:

* contraindications to epidural analgesia
* opioids consumption within the last 24 hours
* patient's unwillingness
* inability to comprehend or comply with the procedure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-11-05 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2018-12-11 (Actual)

PRIMARY OUTCOMES:
satisfaction visual analog scale (SVAS) measurment | procedure
  The degree of satisfaction is assessed using a satisfaction visual analog scale (SVAS) where 0 corresponded to " completely unsatisfied " and 100 to " completely satisfied ".

SECONDARY OUTCOMES:
Number and intensity of motor block | procedure
  Incidence of motor block determined by number and intensity
Number of call of the aneshetist for insufficient analgesia | procedure
  Number of call of the aneshetist for insufficient analgesia
Number of doses of complementary manual bolus | procedure
  Number of doses of complementary manual bolus administered
Obstetrical informations | procedure
  time of the intervention, doses of oxytocin and prostin used, instrumental delivery
Numbers of Adverse events | procedure
  Numbers of Adverse events (Pruritus, nausea / vomitings, episodes of arterial low blood pressure)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick SENGES, MD, Principal Investigator — University Hospital, Limoges
Locations (1):
- Universiy hospital, Limoges, France